CLINICAL TRIAL: NCT05148624
Title: Comparative Study Between Short-time Bed Rest and Immediate Ambulation After Embryo Transfer Procedure. A Randomized Controlled Trial
Brief Title: Immediate Ambulation Versus Short-time Bed Rest in Sub-fertile Women Undergoing Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dubai Fertility Center (Other)
Responsible Party: Principal Investigator, Mohamed Elkalyoubi, Consultant Obs Gyn and reproductive medicine - Head of Medical Affair, Dubai Fertility Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Bed rest after embryo transfer
Record Dates: First submitted 2021-10-15; First posted 2021-12-08 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Infertility, Female
Keywords: Embryo transfer; Bed rest; Clinical pregnancy; Miscarriage; Ongoing pregnancy
MeSH Terms: conditions — Infertility, Female; Abortion, Spontaneous | interventions — Embryo Transfer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate ambulation (Experimental): Sub-infertile women will immediately ambulate and empty her bladder after embryo transfer.
  Interventions: Procedure: embryo transfer
- short time bed rest (Active Comparator): Sub-infertile women will stay in the bed (same bed where embryo transfer was performed) after embryo transfer for a period of 5 minutes without emptying her bladder.
  Interventions: Procedure: embryo transfer

INTERVENTIONS:
Procedure: embryo transfer — immediate ambulation after embryo transfer

SUMMARY:
Bed rest after embryo transfer (ET) has been clinically advised without robust scientific evidence. In investigators' unit, post ET instructions are given immediately after ET to sub-fertile women while lying in bed. The aim of the study is to compare the reproductive outcome of this practice compared with immediate ambulation and giving instructions after emptying the bladder.

DETAILED DESCRIPTION:
Bed rest after embryo transfers has been clinically advised without robust scientific evidence. Most of the assisted reproductive units routinely recommend a variable period of bedrest immediately after embryo transfer (ET) procedure without clear scientific evidence of its benefit. Three Randomized controlled trials (RCT) that included 712 embryo transfers with variable duration of bedrest did not report a benefit in pregnancy outcome. Only one study, however compared bedrest with no bedrest. In contrast, a 2013 RCT reported a harmful effect on the pregnancy outcome.

However, data on patients using embryos derived from their own oocytes are limited. In addition, there was no subgroup analysis to exclude confounding factors like number of oocytes retrieved and quality of embryos transferred. Few of these studies included embryos transferred after preimplantation genetic diagnosis.

The rationale behind bedrest come from the belief that decreased physical activity will help in embryo retention within the uterine cavity after replacement6. Ultrasound examination before and after ET with immediate ambulation did not show any uterine displacement of the air bubble. if gravity displaces transferred embryos, then staying with full bladder in supine position will make the anteverted ante flexed uterus more horizontal and increase the gravity effect.

Moreover, although bed rest is one of the most practiced treatments to improve reproductive outcome, most clinicians consider it the least crucial factor.

In investigators' unit, post ET instructions, which, may take up to 5 minutes, are practiced immediately after ET to patients while lying in bed. The aim of the study is to compare the effect of this practice with immediate ambulation and giving instructions after emptying the bladder in a sitting position on the reproductive outcome in patients undergoing assisted reproductive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Couple undergoing In vitro fertilization, Intracytoplasmic sperm injection, Frozen embryo replacement or Frozen Intracytoplasmic sperm injection
* Age between 20 to 40-year-old
* Couples who are willingly accepting to participate in the study. Both husband and wife will sign the consent.

Exclusion Criteria:

* Women with diminished ovarian reserve (AMH < 1.2 ng/ml or AFC < 7)
* Women with unilateral or bilateral hydro salpinx
* Women with bilateral endometriomas
* Women with adenomyosis
* Women with large (more than 3 cm uterine fibroid)
* Women with fluid or polyp in the uterine cavity
* Women with known chronic endometritis
* Women with H/O recurrent >2 pregnancy loss or implantation failure
* Were enrolled in this study before

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women in reproductive age group who underwent embryo transfer
Enrollment: 156 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who received or did not receive bed rest after embryo transfer who carried a viable pregnancy beyond 10 weeks' gestation | 14 weeks
  Ongoing pregnancy will be defined as a viable pregnancy detected by ultrasound examination between 10 - 13 weeks' gestation.
  The two groups will be compared using relative risk with 95% confidence interval.

SECONDARY OUTCOMES:
Percentage of participants who received or did not receive bed rest after embryo transfer who carried a viable pregnancy beyond 6 weeks' gestation | 6 weeks
  The two groups will be compared using relative risk with 95% confidence interval.
Percentage of participants who received or did not receive bed rest after embryo transfer who aborted before 12 weeks' gestation | 12 weeks
  The two groups will be compared using relative risk with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Cherian, Principal Investigator — Dubai Fertility Center - Dubai Health Authority
Locations (1):
- Dubai Fertility Center, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No